CLINICAL TRIAL: NCT00326391
Title: A Placebo-Controlled, Double-Blind, Parallel-Group, Dose-Titration Study to Evaluate the Efficacy and Safety of CONCERTA (Methylphenidate HCl) Extended-release Tablets in Adults With Attention Deficit Hyperactivity Disorder at Doses of 36 mg, 54 mg, 72 mg, 90 mg, or 108 mg Per Day.
Brief Title: A Safety and Effectiveness Study of Methylphenidate HCl Extended-release Tablets in Adults With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR011560
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity, ADHD, Attention Deficit Disorder Adult
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

INTERVENTIONS:
Drug: methylphenidate hydrochloride extended-release tablets

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of methylphenidate HCl extended-release tablets at five dose levels compared to placebo in adults with Attention Deficit Hyperactivity Disorder (ADHD)

DETAILED DESCRIPTION:
This is a randomized (patients are assigned different treatments based on chance), placebo-controlled , double-blind (neither the patient nor the physician knows whether drug or placebo is being taken), parallel-group, dose-titration, multicenter study to determine the effectiveness and safety of five doses of methylphenidate HCl extended-release tablets, 36 mg, 54 mg, 72 mg (two 36 mg tablets), 90 mg (one 36 mg tablet plus one 54 mg tablet), or 108 mg (two 54 mg tablets) administered orally once per day in adults with Attention Deficit Hyperactivity Disorder. Patients will be randomized to receive either placebo or methylphenidate HCl extended-release tablets for seven weeks. Patients assigned to methylphenidate HCl extended-release tablets will start treatment with 36 mg and continue to receive incremental increases of 18 mg of methylphenidate HCl extended-release tablets every seven days (+/-2 days) until an individualized dose is achieved. The individualized dose is achieved when Adult ADHD Investigator Symptom Rating Scale (AISRS) decreases by 30% and a Clinical Global Impression - Improvement (CGI-I) score is 1 or 2, or titration to the maximum dose of 108 mg is achieved. If a limiting adverse event occurs, the dose will be titrated downward by 18 mg. This dose is then the patient's individualized dose. Once an individualized dose has been achieved, patients will remain on that dose for the duration of the titration period and for the two weeks prior to Final Visit/2-Week Efficacy Assessment Visit. Patients assigned to placebo will follow the same dosing schedule and procedures as the patients randomized to methylphenidate HCl tablets. Safety assessments include monitoring adverse events, blood pressure, pulse, weight, and electrocardiograms (ECG) throughout the study. The primary hypothesis is that methylphenidate HCL extended-release tablets at an individualized dose will be superior to placebo with respect to improvement in the primary efficacy endpoint defined by change from baseline in the Adult ADHD Investigator Symptom Rating Scale. Patients will initiate methylphenidate HCl extended-release tablets with 36 mg and continue to receive increases in 18 mg increments for 7 days until an individualized dose or maximum dose of 108 mg is achieved. Patients will remain on this dose for the duration of the titration period and for 2 weeks prior to Final Visit/2 Week Efficacy Assessment; a maximum of 51 days. Patients receiving placebo will follow the same dosing schedule/procedures as patients receiving methylphenidate HCL tablets

ELIGIBILITY:
Inclusion Criteria:

* Investigator determined diagnosis of ADHD as defined by the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria with symptomatology from childhood to adulthood, symptoms present before age seven years and continue to meet full DSM-IV criteria at time of assessment
* Diagnosis confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) at Baseline and Adult ADHD Investigator Symptom Rating Scale (AISRS) score of 24 or greater as determined by the Investigator at Baseline
* Global Assessment of Functioning (GAF) Scale score of 41 to 60, inclusive, at Baseline
* Minimum weight of 100 lbs (45.4 kg) at Screening
* Negative urine drug test at the Screening and Baseline Visits when tested for drugs of abuse

Exclusion Criteria:

* Known to be non-responders to methylphenidate or other stimulants for the treatment of ADHD
* History of allergy, sensitivity or contraindication to methylphenidate or components of methylphenidate HCL extended-release tablets
* Coexisting medical condition or taking concomitant medication that would interfere with safe administration of methylphenidate in the Investigator's opinion
* Known structural cardiac abnormality
* Diagnosis of or family history of Tourette's syndrome, or motor or verbal tics
* history of seizures or a seizure disorder other than febrile seizures in childhood
* Glaucoma
* Uncontrolled hyperthyroidism or hypothyroidism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The change from Baseline in the Adult ADHD Investigator Symptom Rating Scale (AISRS) total score as assessed by the Investigator at the Final Visit/2 Week Efficacy Assessment Visit

SECONDARY OUTCOMES:
Change from baseline in the AISRS as completed by the Investigator at each Titration Visit. Change from baseline in the AISRS as completed by the Investigator at the end of the study or the last score provided during the study by mg/kg dosing groups.

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Derived] Adler LA, Zimmerman B, Starr HL, Silber S, Palumbo J, Orman C, Spencer T. Efficacy and safety of OROS methylphenidate in adults with attention-deficit/hyperactivity disorder: a randomized, placebo-controlled, double-blind, parallel group, dose-escalation study. J Clin Psychopharmacol. 2009 Jun;29(3):239-47. doi: 10.1097/JCP.0b013e3181a390ce. PMID 19440077
- See also: A Placebo-Controlled, Double-Blind, Parallel-Group, Dose-Titration Study to Evaluate the Efficacy and Safety of CONCERTA� in Adults with Attention Deficit Hyperactivity Disorder at Doses of 36 mg, 54 mg, 72 mg, 90 mg, or 108 mg per day — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1092&filename=CR011560_CSR.pdf